CLINICAL TRIAL: NCT04904744
Title: Effect of Varied Outreach Methods on Appointment Scheduling, Appointment Completion, and Receipt of COVID-19 Vaccination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 2020-0769-1
Record Dates: First submitted 2021-05-25; First posted 2021-05-27 (Actual); Results first posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-08

CONDITIONS: Health Care Utilization; Vaccine Preventable Disease
MeSH Terms: conditions — Patient Acceptance of Health Care; Vaccine-Preventable Diseases | interventions — NMT1 protein, S pombe

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No message (Placebo Comparator): No message sent
  Interventions: Other: No message
- Low tailored message (Active Comparator): 2 text or phone reminders that child is overdue for well child check visit
  Interventions: Other: Low tailored message
- Low tailored message plus COVID-19 vaccine message (Active Comparator): 2 text or phone reminders that child is overdue for well child check visit AND COVID-19 vaccine is available
  Interventions: Other: Low tailored message plus COVID-19 vaccine message

INTERVENTIONS:
Other: Low tailored message — 2 low tailored text or phone message reminders that child is overdue for well child check visit
  Arms: Low tailored message
Other: No message — No reminders are sent
  Arms: No message
Other: Low tailored message plus COVID-19 vaccine message — 2 low tailored text or phone message reminders that child is overdue for well child check visit and that COVID-19 vaccine is available
  Arms: Low tailored message plus COVID-19 vaccine message

SUMMARY:
Our objective is to determine the effectiveness of varied outreach methods to children age 12-17 years old who are due for a well child check visit and don't have one scheduled in the next 45 days on the outcomes of appointment scheduling, appointment completion, and receipt of the COVID-19 vaccination.

ELIGIBILITY:
Inclusion Criteria:

* age 12-17 years
* has not had a well child check in past 365 days
* no future well child check visit scheduled
* parent preferred language = English or Spanish

Exclusion Criteria:

* phone number not available in electronic health record

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1235 (Actual)
Dates: Start 2021-05-28 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Brinkman, MD, Principal Investigator — Cincinnati Children's
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Burkhardt MC, Berset AE, Xu Y, Mescher A, Brinkman WB. Effect of Outreach Messages on Adolescent Well-Child Visits and Coronavirus Disease 2019 Vaccine Rates: A Randomized, Controlled Trial. J Pediatr. 2023 Feb;253:158-164.e1. doi: 10.1016/j.jpeds.2022.09.035. Epub 2022 Oct 4. PMID 36202236

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | No Message | Low Tailored Message | Low Tailored Message Plus COVID-19 Vaccine Message
Started | 412 | 412 | 411
Completed | 412 | 412 | 411
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Message | Low Tailored Message | Low Tailored Message Plus COVID-19 Vaccine Message | Total
Number analyzed (Participants) | 412 | 412 | 411 | 1235
Age, Customized [Number; unit: participants]
  12 | 78 | 74 | 72 | 224
  13 | 99 | 103 | 110 | 312
  14 | 98 | 105 | 106 | 309
  15 | 61 | 57 | 54 | 172
  16 | 33 | 39 | 29 | 101
  17 | 43 | 34 | 40 | 117
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 196 | 192 | 210 | 598
  Male | 216 | 220 | 201 | 637
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 21 | 15 | 51
  Not Hispanic or Latino | 396 | 390 | 396 | 1182
  Unknown or Not Reported | 1 | 1 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 6 | 3 | 2 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 315 | 313 | 319 | 947
  White | 65 | 69 | 60 | 194
  More than one race | 13 | 10 | 17 | 40
  Unknown or Not Reported | 13 | 16 | 13 | 42

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Completed an Adolescent Well-care Visit
Description: Participant completed adolescent well-care visit as determined by the presence of well-visit billing code documented in the electronic health record
Time Frame: Within 8 weeks of the date of intervention or the date of randomization for the control group
Measure: Count of Participants; unit: Participants
Arm/Group | No Message | Low Tailored Message | Low Tailored Message Plus COVID-19 Vaccine Message
Number analyzed (Participants) | 412 | 412 | 411
Participants | 43 | 56 | 55
Statistical Analysis 1: Comparison: No Message vs Low Tailored Message; Test type: Superiority; p = 0.165, Regression, Logistic; Odds Ratio (OR) = 1.35, 95% CI 2-sided [0.88 to 2.06] — Low Tailored Message vs. No Message (reference group)
Statistical Analysis 2: Comparison: No Message vs Low Tailored Message Plus COVID-19 Vaccine Message; Test type: Superiority; p = 0.193, Regression, Logistic; Odds Ratio (OR) = 1.33, 95% CI 2-sided [0.87 to 2.03] — Low tailored message plus COVID-19 vaccine message vs. No Message
Statistical Analysis 3: Comparison: Low Tailored Message vs Low Tailored Message Plus COVID-19 Vaccine Message; Test type: Superiority; p = 0.930, Regression, Logistic; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.68 to 1.52] — Low Tailored Message vs. Low tailored message plus COVID-19 vaccine message

2. Secondary Outcome: Number of Participants Who Scheduled an Adolescent Well-care Appointment
Description: Participant scheduled an adolescent well-care appointment as determined by documentation in electronic health record
Time Frame: Within 2 weeks of the date of intervention or the date of randomization for the control group
Measure: Count of Participants; unit: Participants
Arm/Group | No Message | Low Tailored Message | Low Tailored Message Plus COVID-19 Vaccine Message
Number analyzed (Participants) | 412 | 412 | 411
Participants | 22 | 43 | 27
Statistical Analysis 1: Comparison: No Message vs Low Tailored Message; Test type: Superiority; p = 0.008, Regression, Logistic; Odds Ratio (OR) = 2.07, 95% CI 2-sided [1.21 to 3.52] — Low Tailored Message vs. No Message
Statistical Analysis 2: Comparison: No Message vs Low Tailored Message Plus COVID-19 Vaccine Message; Test type: Superiority; p = 0.457, Regression, Logistic; Odds Ratio (OR) = 1.25, 95% CI 2-sided [0.70 to 2.23] — Low tailored message plus COVID-19 vaccine message vs. No Message
Statistical Analysis 3: Comparison: Low Tailored Message vs Low Tailored Message Plus COVID-19 Vaccine Message; Test type: Superiority; p = 0.049, Regression, Logistic; Odds Ratio (OR) = 1.66, 95% CI 2-sided [1.00 to 2.74] — Low Tailored Message vs. Low tailored message plus COVID-19 vaccine message

3. Secondary Outcome: Participant Receipt of COVID-19 Vaccine
Description: Participant received COVID-19 vaccine as determined by presence of documentation of vaccine administration in the electronic health record.
Time Frame: Within 8 weeks of the date of intervention or the date of randomization for the control group
Measure: Count of Participants; unit: Participants
Arm/Group | No Message | Low Tailored Message | Low Tailored Message Plus COVID-19 Vaccine Message
Number analyzed (Participants) | 412 | 412 | 411
Participants | 8 | 16 | 10
Statistical Analysis 1: Comparison: No Message vs Low Tailored Message; Test type: Superiority; p = 0.104, Regression, Logistic; Odds Ratio (OR) = 2.04, 95% CI 2-sided [0.86 to 4.82] — Low Tailored Message vs. No Message
Statistical Analysis 2: Comparison: No Message vs Low Tailored Message Plus COVID-19 Vaccine Message; Test type: Superiority; p = 0.631, Regression, Logistic; Odds Ratio (OR) = 1.26, 95% CI 2-sided [0.49 to 3.22] — Low tailored message plus COVID-19 vaccine message vs. No Message
Statistical Analysis 3: Comparison: Low Tailored Message vs Low Tailored Message Plus COVID-19 Vaccine Message; Test type: Superiority; p = 0.238, Regression, Logistic; Odds Ratio (OR) = 1.62, 95% CI 2-sided [0.73 to 3.61] — Low Tailored Message vs. Low tailored message plus COVID-19 vaccine message

4. Secondary Outcome: Family Member Receipt of COVID-19 Vaccine
Description: Family member received COVID-19 vaccine as determined by presence of documentation of vaccine administration in the electronic health record.
Time Frame: Within 8 weeks of the date of intervention or the date of randomization for the control group
Population: Data was only available for parents that received a COVID-19 vaccine at one of our academic primary care offices. Thus, information about household members receiving vaccination is likely incomplete due to lack of access to adult medical records and vaccinations administered outside our health system.
Measure: Count of Participants; unit: Participants
Arm/Group | No Message | Low Tailored Message | Low Tailored Message Plus COVID-19 Vaccine Message
Number analyzed (Participants) | 412 | 412 | 411
Participants | 2 | 5 | 3

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | No Message | Low Tailored Message | Low Tailored Message Plus COVID-19 Vaccine Message
All-Cause Mortality (participants affected / at risk) | 0/412 | 0/412 | 0/411
Serious Adverse Events (participants affected / at risk) | 0/412 | 0/412 | 0/411
Other Adverse Events (participants affected / at risk) | 0/412 | 0/412 | 0/411

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-14): https://cdn.clinicaltrials.gov/large-docs/44/NCT04904744/Prot_SAP_000.pdf